CLINICAL TRIAL: NCT01091974
Title: Cognitive Behavioral Therapy +/- Armodafinil for Insomnia and Fatigue Following Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Joseph Roscoe, Research Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: UCCS07090; 1R01CA126968-01A1 (NIH)
Record Dates: First submitted 2009-12-09; First posted 2010-03-24 (Estimated); Results first posted 2015-03-13 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Insomnia; Fatigue; Breast Cancer
Keywords: Insomnia; Fatigue; QOL; CBT; Breast cancer; Survivors; Chemotherapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Fatigue; Breast Neoplasms | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 - CBT-I + placebo (Experimental): CBT-I and placebo
  Interventions: Drug: Placebo Comparator; Behavioral: CBT-I
- 2 - CBT-I + Armodafinil (Experimental): CBT-I + Armodafinil
  Interventions: Drug: armodafinil; Behavioral: CBT-I
- 3 - Placebo only (Placebo Comparator): Placebo only
  Interventions: Drug: Placebo Comparator
- 4 - Armodafinil only (Experimental): Armodafinil only
  Interventions: Drug: armodafinil

INTERVENTIONS:
Drug: armodafinil — Armodafinil P.O. daily/47 days (3-days at 50mg, then 40 days at 100mg, then 4 days at 50mg)
  Arms: 2 - CBT-I + Armodafinil; 4 - Armodafinil only
Drug: Placebo Comparator — Placebo for 47 days
  Arms: 1 - CBT-I + placebo; 3 - Placebo only
Behavioral: CBT-I — Seven weekly sessions of cognitive behavioral therapy for insomnia (CBT-I)
  Arms: 1 - CBT-I + placebo; 2 - CBT-I + Armodafinil

SUMMARY:
This is a four-arm, randomized, controlled, clinical trial examining the efficacy of of cognitive behavioral therapy (CBT)-I and armodafinil in reducing insomnia in 226 female breast cancer patients who report sleep disturbances following completion of chemotherapy.

DETAILED DESCRIPTION:
Treatment Protocol: CBT-I and armodafinil are being studied in a four-arm, randomized, controlled, clinical trial of 226 cancer survivors with chronic insomnia who are at least one month post treatment. The seven-week intervention is designed to determine the efficacy and acceptability of these treatment strategies in reducing insomnia in cancer survivors. Assessments will be made by questionnaires before, during, and two weeks following the study intervention. All ancillary treatments, as appropriate for control of symptoms caused by the cancer or its treatment may be administered as clinically indicated.

Withdrawal of Sleep Medications: All participants, prior to beginning the baseline data collection phase of the study, must have withdrawn from all sleep medications, including: prescription, over-the-counter, CAM and herbal remedies for at least one week prior to beginning the study.

CBT-I (Arms 3 & 4): CBT-I will be provided on an individual basis to all patients in study Arms 3 & 4 by a licensed clinical psychologist trained in CBT-I by Dr. Perlis. Subjects in these two study arms will receive 7 weeks of CBT-I, using a structured research grade protocol developed at the UR-SNRL. This manualized intervention, which exists as a published text: Perlis et al., 2005, includes four essential components: Sleep Restriction Therapy, Stimulus Control Instruction, Sleep Hygiene Guidelines, and a session of cognitive therapy.

Data Collection: Patients will complete the Insomnia Severity (ISI) at the time of consent and every Friday during weeks 3-11 of the study. A follow-up call by study personnel will be made to each participant not currently receiving CBT-I on each of these Fridays to promote compliance, prompt completion, assess potential side effects of study medication, and answer patient questions.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of cancer.
2. Be able to understand written and spoken English
3. Be able to swallow medication
4. Have preferred sleep phase between 7:30 pm and 11:00 am
5. Be willing to discontinue any medications/OTCs/Herbals for sleep for the 11-week study period
6. Be presumed to be in a state of cancer remission; use of tamoxifen, an aromatase inhibitor, and/or Herceptin is permitted
7. Self-report problems with insomnia for at least three months and that the insomnia began or got worse with the onset of cancer or treatment
8. Have completed chemotherapy and or radiation not less than one month ago. Note: Both types of treatment must be completed at least one month ago if patient receives chemotherapy and radiation therapy and there is no outer limit to how long ago treatments were completed.)
9. Report insomnia on the SDS-CL at a frequency of at least 3 days a week

Exclusion Criteria:

1. Have ever taken modafinil or had CBT-I therapy. CBT-I therapy for the sake of this protocol will be defined as any cognitive behavioral-based treatment for insomnia that includes a sleep restriction component.
2. Have an unstable medical or psychiatric illness (Axis I-current or within the last 5 years)
3. Have a history of seizures or severe headaches, or uncontrolled cardiac disease or hypertension
4. Be presently taking an anticoagulant or a corticosteroid
5. Have taken amphetamines (e.g., methylphenidate, pemoline [Cylert®] or similar psycho stimulants) within the past 30 days
6. Be currently pregnant or nursing
7. Have a history of substance abuse, or meet criteria for current alcohol abuse or dependence as assessed by a CAGE test score >=2 or an Alcohol Use Disorders Identification Test (AUDIT) score >=13
8. Have surgery planned within the study period
9. Have have ever been diagnosed with sleep apnea or have sleep apnea as indicated by endorsing either question 11 (I wake up choking or gasping for air) or question 12 (My bed partner has noticed that I seem to stop breathing) on the Sleep Disorders Symptom Check at the "Often" or "Frequently" level.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2008-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Roscoe, PhD, Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - University of Rochester James P. Wilmot Cancer Center, Rochester, New York
  - Behavioral Sleep Medicine Program, Department of Psychiatry, University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811
- [Derived] Peoples AR, Garland SN, Pigeon WR, Perlis ML, Wolf JR, Heffner KL, Mustian KM, Heckler CE, Peppone LJ, Kamen CS, Morrow GR, Roscoe JA. Cognitive Behavioral Therapy for Insomnia Reduces Depression in Cancer Survivors. J Clin Sleep Med. 2019 Jan 15;15(1):129-137. doi: 10.5664/jcsm.7586. PMID 30621831
- [Derived] Roscoe JA, Garland SN, Heckler CE, Perlis ML, Peoples AR, Shayne M, Savard J, Daniels NP, Morrow GR. Randomized placebo-controlled trial of cognitive behavioral therapy and armodafinil for insomnia after cancer treatment. J Clin Oncol. 2015 Jan 10;33(2):165-71. doi: 10.1200/JCO.2014.57.6769. Epub 2014 Dec 1. PMID 25452447

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 138 Patients were consented of which 114 were eligible.
Pre-assignment Details: 18 Withdrew prior to randomization (3 ceased responding to contacts, 4 changed mind , 3 began or restarted sleep medication, 4 did not complete baseline measures, 1 did not receive approval from physician to participate, 1 found the diaries too much trouble, 1 did not want to take study medication, and 1 had a family emergency).
Groups:
- Arm 1 - (CBT-I) + Placebo: Placebo Comparator: Placebo for 47 days
  CBT-I: Seven weekly sessions of cognitive behavioral therapy for insomnia (CBT-I)
- 3- Placebo Only: Placebo Comparator: Placebo for 47 days
Period: Overall Study
Arm/Group | Arm 1 - (CBT-I) + Placebo | 2 - CBT-I + Armodafinil | 3- Placebo Only | 4 - Armodafinil Only
Started | 24 | 23 | 25 | 24
Completed | 19 | 18 | 19 | 17
Not Completed | 5 | 5 | 6 | 7
Not completed — Did not start intervention | 3 | 1 | 3 | 1
Not completed — resumed sleep medication | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 3 | 2 | 2
Not completed — side-effects | 1 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 - CBT-I + Placebo | 2 - CBT-I + Armodafinil | 3 - Placebo Only | 4 - Armodafinil Only | Total
Number analyzed (Participants) | 24 | 23 | 25 | 24 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (9.9) | 56 (10.2) | 52 (11.5) | 57 (7.4) | 56.1 (10.0)
Gender [Count of Participants; unit: Participants]
  Female | 21 | 22 | 18 | 23 | 84
  Male | 3 | 1 | 7 | 1 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 22 | 24 | 22 | 91
  Unknown or Not Reported | 1 | 1 | 1 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 4 | 1 | 8
  White | 23 | 21 | 19 | 23 | 86
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 24 | 23 | 25 | 24 | 96

OUTCOME MEASURES:

1. Primary Outcome: Change in Insomnia Severity Index From Baseline to Post-intervention
Description: The Insomnia Severity Index (ISI) is a commonly used, 7-item psychometrically validated measure used to rate insomnia with 0-7 = absence of insomnia, 8-14 = subthreshold insomnia symptoms, 15-21 = moderate insomnia, and 22-28 = severe insomnia.
Time Frame: ANCOVA was employed with multiple imputation on the post-intervention score (average of the two post-intervention weeks), controlling for the score at the time of consent (pre).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1 - (CBT-I) + Placebo | 2 - CBT-I + Armodafinil | 3- Placebo Only | 4 - Armodafinil Only
Number analyzed (Participants) | 24 | 23 | 25 | 24
units on a scale | -4.93 (1.85) | -6.36 (1.84) | 1.04 (1.89) | -1.43 (1.78)

2. Secondary Outcome: Fatigue Will be Assessed by the Total Score of the Revised Brief Fatigue Inventory (BFI) .
Description: The revised Brief Fatigue Inventory (BFI) is a 9-item, patient-report instrument with established reliability and validity. The BFI allows for the rapid assessment of fatigue level in cancer patients and identifies those patients with severe fatigue. Three items ask patients to rate their fatigue "now," and fatigue at its "worst" and "usual" for the last 24 hours. The 11-point scales are bounded by 0 = "no fatigue" and 10 = "fatigue as bad as you can imagine." Using the same type of scales, the remaining questions ask patients to rate how their fatigue interferes with several functional domains, including general activity, walking, mood, work, and relations with others. These scales are bounded by 0 = "does not interfere" and 10 = "interferes completely." A global fatigue score (ranging from 0-10) can be obtained by averaging all the items on the BFI.
Time Frame: as for outcome 1
Population: Note: One patient randomized to the placebo only condition failed to provide data and was not included in the analyses.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1 - (CBT-I) + Placebo | 2 - CBT-I + Armodafinil | 3- Placebo Only | 4 - Armodafinil Only
Number analyzed (Participants) | 24 | 23 | 24 | 24
units on a scale | 2.041 (0.411) | 1.209 (0.364) | 2.971 (0.534) | 3.167 (0.456)

ADVERSE EVENTS:
Time Frame: Participants were followed throughout the study duration, for up to 24 weeks
Arm/Group | Arm 1 - (CBT-I) + Placebo | 2 - CBT-I + Armodafinil | 3- Placebo Only | 4 - Armodafinil Only
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 3/23 | 0/25 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - (CBT-I) + Placebo (N=24) | 2 - CBT-I + Armodafinil (N=23) | 3- Placebo Only (N=25) | 4 - Armodafinil Only (N=24)
Headache (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Numbness/tingling (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes